CLINICAL TRIAL: NCT01695135
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Study of Abiraterone Acetate (JNJ-212082) Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Docetaxel-Based Chemotherapy
Brief Title: A Study of Abiraterone Acetate Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer Who Have Failed Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100010; ABI-PRO-3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-05

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Metastatic castration resistant prostate cancer; Abiraterone acetate; JNJ-212082
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abiraterone acetate plus prednisone (Experimental)
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone
- Placebo plus prednisone (Experimental)
  Interventions: Drug: Placebo; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone 1000 mg (4 x 250 mg tablets) taken orally once daily
  Arms: Abiraterone acetate plus prednisone
Drug: Placebo — Placebo (4 tablets) taken orally once daily
  Arms: Placebo plus prednisone
Drug: Prednisone — Prednisone 5 mg tablet taken orally twice daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of abiraterone acetate when co-administered with prednisone in Asian patients with metastatic castration-resistant prostate cancer (mCRPC) who have failed docetaxel-based chemotherapy.

DETAILED DESCRIPTION:
This is a randomized (the treatment group is assigned by chance), double-blind (neither physician nor patient knows the treatment that the patient receives) placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study with a randomization allocation ratio of 2:1 between the abiraterone acetate group (abiraterone acetate plus prednisone) and the placebo group (placebo plus prednisone). Approximately 200 (133 in the abiraterone acetate group and 67 in the placebo group) medically or surgically castrated male patients with mCRPC who have failed docetaxel-based chemotherapy will be enrolled in this study for up to 27 months. The study protocol includes the following phases: screening (within 28 days prior to randomization on Cycle 1 Day 1), double-blind treatment (28-day cycles until protocol-defined disease progression or unacceptable toxicity), and survival follow-up (up to Month 60). During the follow-up phase, patients with disease progression will be provided open-label (identity of assigned study drug will be known) extension treatment with abiraterone acetate. In the event of a positive study result at the time of the final analysis, participants in the placebo group who have not shown progressive disease in the double-blind treatment Phase of the study will be enrolled in an open-label extension treatment with abiraterone acetate treatment based on the participant's choice and treating physician's endorsement if they meet the criteria for subsequent abiraterone acetate. Abiraterone acetate 1000 mg tablets or placebo will be taken orally (by mouth) once daily plus prednisone 5 mg tablet orally twice daily. Efficacy and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate except neuroendocrine carcinoma including small cell carcinoma
* Disease progressed on or after prior docetaxel-containing chemotherapy
* Prior 1 or 2 cytotoxic chemotherapy regimens for metastatic castration-resistant prostate cancer, at least 1 of which contains docetaxel
* Documented prostate cancer progression as documented by prostate specific antigen progression according to Prostate Specific Antigen Working Group criteria or radiographic progression in soft tissue or bone
* Surgically or medically castrated, with serum testosterone level <50 ng/dL (1.7 nmol/L)
* Eastern Cooperative Oncology Group performance status score of <=2
* Protocol-defined laboratory values
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone (corticosteroid) use contraindicated
* Any chronic medical condition requiring a higher dose of corticosteroid than 5 mg prednisone twice daily
* Pathological finding consistent with neuroendocrine carcinoma of prostate including small cell carcinoma
* Uncontrolled hypertension (systolic BP >=160 mmHg or diastolic BP >=95 mmHg; patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy)
* Active or symptomatic viral hepatitis or chronic liver disease, have a known infection with human immunodeficiency virus and/or hepatitis B virus or hepatitis C virus
* History of pituitary or adrenal dysfunction.
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association Class III or IV heart disease or cardiac ejection fraction measurement of <50% at baseline
* Atrial fibrillation, or other cardiac arrhythmia requiring therapy
* Other malignancy within past 3 years (except basal or nonmetastatic squamous cell carcinoma of the skin)
* Known brain metastasis
* Prior therapy with abiraterone acetate or other CYP17 inhibitor(s), or investigational agent(s) targeting the androgen receptor for metastatic prostate cancer
* Prior therapy with ketoconazole for prostate cancer
* Surgery or local prostatic intervention within 30 days of the first dose
* Radiotherapy, chemotherapy, or immunotherapy within 30 days, or single fraction of palliative radiotherapy within 14 days of administration of Cycle 1 Day 1
* Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a National Cancer Institute-Common Terminology Criteria for Adverse Events grade of <=1 (chemotherapy induced alopecia and grade 2 peripheral neuropathy is allowed)
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of Cycle 1 Day 1
* Anti-androgen treatment must not be given within 4 weeks (flutamide) or 6 weeks (bicalutamide or nilutamide) prior to Cycle 1 Day 1
* Prior systemic treatment with an azole drug (eg, fluconazole, itraconazole) within 4 weeks prior to Cycle 1 Day 1
* Has known allergies, hypersensitivity, or intolerance to abiraterone acetate or its excipients
* Has contraindications to the use of prednisone per local prescribing information
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- China (11):
  - Beijing
  - Changsha
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Tianjin
  - Wenzhou
  - Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 214 participants were enrolled in the study (143 participants in abiraterone acetate group and 71 participants in placebo group).
Groups:
- Placebo + Prednisone (Double-blind [DB]): Participants received placebo (4 tablets) once daily + prednisone 5 milligram (mg) twice daily on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Each cycle of 28 days.
- Abiraterone Acetate + Prednisone (Double-blind): Participants received abiraterone acetate (AA) 1000 mg (4*250 mg tablets) once daily + prednisone 5 mg twice daily on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Each cycle of 28 days.
- Placebo + Prednisone (DB) to AA + Prednisone (Open-label); AA + Prednisone to AA + Prednisone (Open-label): Participants with disease progression during the double-blind treatment phase received abiraterone acetate 1000 mg once daily + prednisone 5 mg twice daily in open-label extension treatment phase based on the participant's choice and treating physician's decision if they met the criteria for subsequent abiraterone acetate treatment until they no longer derive clinical benefit, unacceptable toxicity, initiation of a subsequent anticancer therapy, or serious protocol violation.
Period: Double-blind Treatment Phase
Arm/Group | Placebo + Prednisone (Double-blind [DB]) | Abiraterone Acetate + Prednisone (Double-blind) | Placebo + Prednisone (DB) to AA + Prednisone (Open-label) | AA + Prednisone to AA + Prednisone (Open-label)
Started | 71 | 143 | 0 | 0
Completed | 0 | 4 | 0 | 0
Not Completed | 71 | 139 | 0 | 0
Not completed — Progressive disease | 50 | 110 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 14 | 0 | 0
Not completed — Adverse Event | 7 | 7 | 0 | 0
Not completed — Other | 1 | 3 | 0 | 0
Not completed — Physician Decision | 6 | 3 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Noncompliance with study drug | 0 | 1 | 0 | 0
Period: Open Label Extension Treatment Phase
Arm/Group | Placebo + Prednisone (Double-blind [DB]) | Abiraterone Acetate + Prednisone (Double-blind) | Placebo + Prednisone (DB) to AA + Prednisone (Open-label) | AA + Prednisone to AA + Prednisone (Open-label)
Started | 0 | 0 | 49 | 80
Completed | 0 | 0 | 9 | 10
Not Completed | 0 | 0 | 40 | 70
Not completed — Progressive disease | 0 | 0 | 13 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 16
Not completed — Adverse Event | 0 | 0 | 11 | 16
Not completed — Other | 0 | 0 | 4 | 7
Not completed — Physician Decision | 0 | 0 | 4 | 1
Not completed — Death | 0 | 0 | 2 | 7
Not completed — Noncompliance with study drug | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Prednisone (Double-blind): Participants received placebo (4 tablets) once daily + prednisone 5 milligram (mg) twice daily on Cycle 1 Day 1 until disease progression or unacceptable toxicity. Each cycle of 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind) | Total
Number analyzed (Participants) | 71 | 143 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.75) | 68.2 (8.3) | 68 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 71 | 143 | 214
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 71 | 143 | 214
Region of Enrollment [Count of Participants; unit: Participants]
  China | 71 | 143 | 214

OUTCOME MEASURES:

1. Primary Outcome: DB Phase: Time to Prostate-Specific Antigen Progression (PSA)
Description: Time to PSA progression was defined as time interval from the date of randomization to the date of the prostate-specific antigen (PSA) progression as defined in the Prostate Specific Antigen Working Group (PSAWG) criteria. PSAWG criteria- Decline from baseline and reach response criteria: greater than or equal to (>=) 50 percent (%) increase over the nadir and the increase in the absolute-value by at least 5 nanogram per milliliter (ng/mL) (or back to the baseline), which is confirmed by a second value 4 or more weeks later; Decline from baseline but not reach response criteria: >=25% increase over the nadir and the increase in the absolute-value by at least 5 ng/mL, which is confirmed by a second value 4 or more weeks later; and No decline from baseline: >=25% increase over the baseline and the increase in the absolute-value by at least 5 ng/mL, which is confirmed by a second value 4 or more weeks later.
Time Frame: Up to 1.8 years
Population: Intent-to-Treat (ITT) analysis set included all participants randomized into the study and classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 71 | 143
Days | 84.00 [31.00 to 113.00] | 169.00 [141.00 to 197.00]
Statistical Analysis 1: Comparison: Placebo + Prednisone (Double-blind) vs Abiraterone Acetate + Prednisone (Double-blind); Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.528, 95% CI 2-sided [0.376 to 0.740]

2. Secondary Outcome: DB Phase: Overall Survival
Description: Overall survival was defined as the time interval from the date of randomization to the date of death from any cause.
Time Frame: From randomization to the date of death due to any cause (up to approximately 3.8 years)
Population: ITT analysis set included all participants randomized into the study and classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 71 | 143
Days | 561.00 [352.00 to 787.00] | 579.00 [504.00 to 731.00]

3. Secondary Outcome: DB Phase: Percentage of Participants Who Achieved PSA Response
Description: Percentage of participants who achieved PSA response (defined as >= 50% PSA decline from baseline) according to PSAWG criteria were reported. PSAWG criteria- Decline from baseline and reach response criteria: >= 50% increase over the nadir and the increase in the absolute-value by at least 5 ng/mL (or back to the baseline), which is confirmed by a second value 4 or more weeks later; Decline from baseline but not reach response criteria: >=25% increase over the nadir and the increase in the absolute-value by at least 5 ng/mL, which is confirmed by a second value 4 or more weeks later; and No decline from baseline: >=25% increase over the baseline and the increase in the absolute-value by at least 5 ng/mL, which is confirmed by a second value 4 or more weeks later.
Time Frame: Approximately up to 3.8 years
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 71 | 143
Percentage of Participants | 18.3 | 54.5

4. Secondary Outcome: DB Phase: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with measurable disease at baseline achieving a complete response (CR) or partial response (PR) according to modified response evaluation criteria in solid tumors (RECIST) criteria. RECIST criteria for CR: disappearance of all target lesions and non-target lesions and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Approximately up to 3.8 years
Population: ITT analysis set included all participants randomized into the study and classified according to their assigned treatment group, regardless of the actual treatment received. Population included only participants with measurable disease at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 24 | 57
Percentage of Participants | 4.2 | 17.5

5. Secondary Outcome: DB Phase: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Questionnaire: Total Scores at the End of Treatment
Description: FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS) (Range 1-156, higher scores better). The FACT-General (FACT-G) is a 28 item Quality of Life (QOL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional (0-24) Well-being. The total range was between 1-108, higher scores better. Functional Assessment of Cancer Therapy-Treatment Outcome Index (FACT-TOI) is derived from the sum of the Physical Well-Being, Functional Well-Being, and Prostate Cancer subscale scores; a sensitive measure of patient-reported health (Range 1-104, higher scores better). PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better).
Time Frame: Baseline, at End of Treatment (15 and 30 days after the last dose [up to 3.8 years])
Population: ITT analysis set included all participants randomized into the study and classified according to their assigned treatment group, regardless of the actual treatment received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 52 | 97
Units on a scale
  Total Score | -19.9 (22.07) | -16.1 (22.74)
  Physical Well-being | -6.7 (6.52) | -4.9 (6.85)
  Functional Well-being | -5.1 (6.60) | -2.7 (7.31)
  Emotional Well-being | -2.1 (4.48) | -2.4 (4.87)
  Social Well-being | -0.8 (3.82) | -1.2 (6.55)
  FACT-G Total Score | -14.6 (16.25) | -11.2 (17.19)
  Prostate Cancer Subscale (PCS) | -5.3 (7.99) | -4.9 (7.70)
  Treatment Outcome Index (FACT-TOI) | -17.1 (17.76) | -12.5 (17.52)

6. Secondary Outcome: DB Phase: Time to Pain Progression
Description: Time to Pain progression calculated as number of days from date of randomization to date of pain progression. Pain progression- worsening of pain due to metastatic bone disease defined as increase of >=30% in worst pain over past 24 hours on BPI-SF numeric rating scale at 2 consecutive evaluations 4 weeks apart without decrease in analgesic usage score (in 2 corresponding consecutive evaluation in analgesic usage score, if there is missing visit, use existing visit only) or increase in analgesic usage score >=30% at 2 consecutive evaluations 4 weeks apart. BPI-SF is 11-item questionnaire which includes 4 questions that assess pain intensity and 7 questions that assess impact of pain on daily functions. Total score (average of individual questions) ranges from 0=No pain to 10=Pain as bad as you can imagine; Higher scores= greater pain. Analgesic usage was scored on scale of 0 to 3 where 0=no analgesic, 1=non-opioid analgesics, 2=opioids for moderate pain and 3=opioids for severe pain.
Time Frame: Approximately up to 3.8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 71 | 143
Days | 169.00 [85.00 to 253.00] | 505.00 [365.00 to NA] — Here 'NA' represents that upper limit of Confidence Interval (CI) was not estimable due to lesser number of events.

7. Secondary Outcome: DB Phase: Percentage of Participants Experiencing Pain Palliation
Description: Percentage of participants experiencing pain palliation were reported. A participant is responder if experienced >=30% reduction in Brief Pain Inventory - Short Form (BPI-SF) worst pain intensity score over 24 hours observed at 2 consecutive evaluations 4 weeks apart without any increase in analgesic usage score (best response). Analgesic usage was scored on a scale of 0 to 3 where 0=no analgesic, 1=non-opioid analgesics, 2=opioids for moderate pain and 3=opioids for severe pain. BPI-SF is 11-item self-reported questionnaire designed to assess severity and impact of pain on daily functions. It includes 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Total score (average of individual questions) ranges from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Approximately up to 3.8 years
Population: ITT analysis set included all participants randomized into the study and classified according to their assigned treatment group, regardless of the actual treatment received. Population included only participants whose pain score was >= 4 at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 22 | 55
Percentage of Participants | 31.8 | 54.5

8. Secondary Outcome: DB Phase: Change From Baseline in Brief Fatigue Inventory (BFI) Score at End of Treatment
Description: The Brief Fatigue Inventory (BFI) is a brief participant-reported questionnaire that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. BFI has nine items. Three items ask patients to rate the severity of their fatigue at its "worst," "usual," and "now" during normal waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." Six items assess the amount that fatigue has interfered with different aspects of the patient's life during the past 24 hours. The interference items include general activity, mood, walking ability, normal work (includes both work outside the home and housework), relations with other people, and enjoyment of life. The interference items are measured on a 0-10 scale, with 0 being "does not interfere" and 10 being "completely interferes." BFI Total Score is the average of the nine items, ranging from 0 (no fatigue) to 10 (high fatigue).
Time Frame: Baseline, at End of Treatment (15 and 30 days after the last dose [up to 3.8 years])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind)
Number analyzed (Participants) | 52 | 98
Units on a scale
  Fatigue Now | 2.4 (3.59) | 1.7 (3.34)
  Usual Fatigue | 2.4 (3.53) | 1.5 (3.18)
  Worst Fatigue | 2.6 (3.73) | 1.6 (3.49)
  General Activity | 2.3 (3.65) | 1.7 (3.38)
  Mood | 2.7 (3.39) | 1.8 (3.40)
  Walking Ability | 2.4 (3.28) | 1.8 (3.50)
  Normal Work | 2.2 (3.84) | 2.0 (3.71)
  Relations with Other People | 2.0 (3.08) | 1.6 (3.25)
  Enjoyment of Life | 2.5 (3.33) | 1.9 (3.64)

ADVERSE EVENTS:
Time Frame: Approximately up to 3.8 years
Description: Safety analysis set included all randomized participants who received at least one dose of study drug and classified to the treatment group according to their actual treatment received.
Arm/Group | Placebo + Prednisone (Double-blind) | Abiraterone Acetate + Prednisone (Double-blind) | Placebo + Prednisone (DB) to AA + Prednisone (Open-label) | AA + Prednisone to AA + Prednisone (Open-label)
Serious Adverse Events (participants affected / at risk) | 20/71 | 33/143 | 25/49 | 41/80
Other Adverse Events (participants affected / at risk) | 62/71 | 134/143 | 35/49 | 54/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone (Double-blind) (N=71) | Abiraterone Acetate + Prednisone (Double-blind) (N=143) | Placebo + Prednisone (DB) to AA + Prednisone (Open-label) (N=49) | AA + Prednisone to AA + Prednisone (Open-label) (N=80)
Disease progression (General disorders) | 5 | 6 | 8 | 17
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 2 | 3
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 4
Death (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 2 | 3 | 4
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1 | 0 | 1
Viith nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhagic infarction (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone (Double-blind) (N=71) | Abiraterone Acetate + Prednisone (Double-blind) (N=143) | Placebo + Prednisone (DB) to AA + Prednisone (Open-label) (N=49) | AA + Prednisone to AA + Prednisone (Open-label) (N=80)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 36 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 20 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 17 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 17 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 10 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 12 | 29 | 7 | 9
Alanine aminotransferase increased (Investigations) | 9 | 20 | 6 | 5
Blood lactate dehydrogenase increased (Investigations) | 6 | 10 | 3 | 3
Blood albumin decreased (Investigations) | 4 | 8 | 0 | 2
Weight decreased (Investigations) | 3 | 8 | 3 | 9
Blood alkaline phosphatase increased (Investigations) | 6 | 6 | 2 | 3
Platelet count decreased (Investigations) | 2 | 6 | 4 | 6
White blood cell count decreased (Investigations) | 3 | 3 | 4 | 3
Blood phosphorus decreased (Investigations) | 0 | 2 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 2 | 7
White blood cells urine positive (Investigations) | 0 | 1 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 39 | 8 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 17 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 9 | 3 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 3 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 16 | 38 | 13 | 29
Fatigue (General disorders) | 5 | 13 | 1 | 1
Pyrexia (General disorders) | 3 | 12 | 3 | 5
Oedema peripheral (General disorders) | 9 | 10 | 2 | 5
Pain (General disorders) | 4 | 1 | 0 | 0
Hypertension (Vascular disorders) | 9 | 22 | 3 | 4
Urinary tract infection (Infections and infestations) | 6 | 13 | 6 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 10 | 4 | 4
Constipation (Gastrointestinal disorders) | 5 | 12 | 2 | 4
Nausea (Gastrointestinal disorders) | 3 | 5 | 1 | 4
Vomiting (Gastrointestinal disorders) | 6 | 4 | 3 | 3
Haematuria (Renal and urinary disorders) | 4 | 9 | 2 | 1
Proteinuria (Renal and urinary disorders) | 5 | 9 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 9 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 3 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 5 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.